CLINICAL TRIAL: NCT06133114
Title: Psychopharmacological Treatment of Emotional Distress: A Randomized Controlled Trial
Brief Title: Psychopharmacological Treatment of Emotional Distress
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Igor Galynker, Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01296
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Suicide Crisis Syndrome; Psychological Distress
MeSH Terms: interventions — Clonazepam; Olanzapine; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- S arm: Single drug clonazepam (Experimental): Single drug clonazepam: 1 mg a day (0.5 mg twice a day) with Treatment As Usual (TAU)
  Interventions: Drug: Clonazepam
- D arm: Two-drug combination clonazepam/olanzapine (Experimental): Two-drug combination clonazepam/olanzapine: 1 mg a day (0.5 mg twice a day) of Clonazepam plus 2.5 mg a day of Olanzapine with Treatment As Usual (TAU)
  Interventions: Drug: Clonazepam; Drug: Olanzapine
- T arm: Three-drug combination clonazepam/olanzapine/buprenorphine (Experimental): Three-drug combination clonazepam/olanzapine/buprenorphine: 1 mg a day (0.5 mg twice a day) of Clonazepam plus 2.5 mg a day of Olanzapine plus 2mg a day of Buprenorphine with Treatment As Usual (TAU)
  Interventions: Drug: Clonazepam; Drug: Olanzapine; Drug: Buprenorphine
- Control Group (No Intervention): Participants that will not receive an intervention.

INTERVENTIONS:
Drug: Clonazepam — 0.5 mg twice a day (1 mg a day)
  Other Names: TAU
  Arms: D arm: Two-drug combination clonazepam/olanzapine; S arm: Single drug clonazepam; T arm: Three-drug combination clonazepam/olanzapine/buprenorphine
Drug: Olanzapine — 2.5 mg once a day of Olanzapine
  Arms: D arm: Two-drug combination clonazepam/olanzapine; T arm: Three-drug combination clonazepam/olanzapine/buprenorphine
Drug: Buprenorphine — 2 mg once a day of Buprenorphine
  Arms: T arm: Three-drug combination clonazepam/olanzapine/buprenorphine

SUMMARY:
This is an inpatient four-arm randomized control trial comparing single drug clonazepam (S arm), a two-drug combination clonazepam/olanzapine (D arm), and a three-drug combination clonazepam/olanzapine/buprenorphine (T arm) with treatment as usual (TAU arm) in the treatment of emotional distress, specifically the Suicide Crisis Syndrome (SCS). All participants in experimental arms receive 2-day pulse treatments targeting four out of five of the acute emotional distress symptoms. The primary outcome measure is SCS at discharge and one-month follow-up. The secondary outcome measures include questions about suicidal behaviors associated with emotional distress at a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to an inpatient unit and ruled in for SCS diagnosis using SCS-C
* Willing to stay in the hospital voluntarily, if medically necessary, for at least 4 days after enrolling in the study.
* Patient admitted to an inpatient unit as a result of a recent (i.e., past-month) suicide attempt, as defined by the C-SSRS (Columbia Suicide Rating Scale).
* Admitted to an inpatient unit in the last 36 hrs.
* Able to understand the nature and the substance of the consent form.
* Currently domiciled.
* Able and willing to provide verifiable contact information for follow-up.

Exclusion Criteria:

* Intellectual disability, cognitive impairment, or linguistic limitation precluding understanding of the consent or research questions.
* Past adverse reactions to clonazepam, olanzapine, or buprenorphine
* Past history of opiate or benzodiazepine use d/o in the last 2 years
* On agonist therapy for opiate addiction
* Ongoing treatment with clonazepam or olanzapine.
* Significant medical or neurological disease or possible delirium that might interfere with study participation or capacity to provide informed consent.
* Receiving involuntary treatment in psychiatric unit
* Clinical suspicion of malingering by a CP.
* Undomiciled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Suicide Crisis Syndrome-Checklist (SCS-C) | up to 1 month follow up after discharge
  The SCS-C is a clinician rated measure assessing clinicians' assessment of the presence and intensity of the Suicide Crisis Syndrome among their patients. The SCS-C includes 13 dichotomous items reflecting the presence or absence of the SCS symptoms. The SCS-C also assesses the presence of the five SCS criteria (entrapment, affective disturbances, loss of cognitive control, hyperarousal and social withdrawal). The first item is a clinician rating of entrapment (SCS criterion A), rated as yes or no. The second item assesses the 4 domains of SCS criterion B: affective disturbance, loss of cognitive control, hyperarousal, and social withdrawal.
  This item is rated yes if the patient exhibits 1 of the domains. A final rating is recorded as positive if both criteria A and B are rated as yes. A positive rating in the final rating reflects a positive SCS diagnosis.

SECONDARY OUTCOMES:
Suicide Crisis Inventory-Short Form (SCI-SF) for Severity | up to 1 month follow up after discharge
  The SCI-SF is an 8-item version of the original 49-item Suicide Crisis Inventory that assesses the severity of different cognitive and affective states theorized in the SCS. Patients rate how they feel on a 5-point scale ranging from 0 (not at all) to 4 (extremely), with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Galynker, MD,PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigator in individual journals.